CLINICAL TRIAL: NCT00338273
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Aripiprazole in the Treatment of Patients With Bipolar I Disorder With a Major Depressive Episode
Brief Title: A Study of Aripiprazole in Patients With Bipolar I Disorder With a Major Depressive Episode
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-149
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2012-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I disorder with major depressive episode
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 5 - 30 mg, Once daily, 8 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, 0 mg, Once daily, 8 weeks.
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate flexible doses (5-30 mg) of aripiprazole in patients with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Must sign informed consent prior to protocol-related procedures

Exclusion Criteria:

* Women who are pregnant, trying to become pregnant, or nursing
* Significant risk of committing suicide
* Any serious unstable medical conditions

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint (Week 8 last observation carried forward = LOCF) on the Montgomery-Asberg Depression Rating Scale (MADRS) total score

SECONDARY OUTCOMES:
Mean change from baseline to endpoint on the Clinical Global Impression-Bipolar Version, severity of illness score (depression)

CONTACTS AND LOCATIONS:
Locations (8):
- Local Institution, Durham, North Carolina, United States
- India (7):
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Chennai
  - Local Institution, Delhi
  - Local Institution, Hyderabad
  - Local Institution, Lucknow
  - Local Institution, Mumbai
  - Local Institution, Visakhapatnam